CLINICAL TRIAL: NCT02373254
Title: Pain Management With NSAIDS in Acute Ankle Fractures Type Supination, External Rotation (SER) II: A Prospective Randomized, Single Blinded Controlled Study
Brief Title: NSAIDS Versus Opioids in Acute SER II Ankle Fractures
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 656916
Record Dates: First submitted 2015-02-09; First posted 2015-02-26 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Ankle Fracture
MeSH Terms: conditions — Ankle Fractures | interventions — Ibuprofen; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ibuprofen 400 mg (Active Comparator): Ibuprofen 400 mg po q 8 hours as needed (PRN) for pain. Subjects will receive Norco, 5/525 mg po q 6 hours PRN if pain relief with Ibuprofen is not sufficient.
  Interventions: Drug: Ibuprofen
- Ibuprofen 800 mg (Active Comparator): Ibuprofen 800 mg po q 8 hours PRN pain. Subjects will receive Norco, 5/525 mg po q 6 hours PRN if pain relief with Ibuprofen is not sufficient.
  Interventions: Drug: Ibuprofen
- Norco (Active Comparator): Norco (acetaminophen/hydrocodone) 10/325 mg po q 6 hours PRN pain. If pain is not relieved, physician should be contacted.
  Interventions: Drug: Acetaminophen/hydrocodone

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen 400 mg and 800 mg
  Other Names: Motrin
  Arms: Ibuprofen 400 mg; Ibuprofen 800 mg
Drug: Acetaminophen/hydrocodone — Norco 5/325 mg and 10/325 mg
  Other Names: Norco
  Arms: Norco

SUMMARY:
This study is being conducted to evaluate whether NSAIDS are more or less effective in bone healing than opioids in acute fracture pain. Participants will be randomized to one of three groups for first line treatment of pain related to the fracture.

DETAILED DESCRIPTION:
Pain management in acute fractures is challenging and influenced by several factors contributing to pain perception. These factors include but are not limited to tissue damage by the local impact, mechanical stress at the fracture ends, and central perception of the noxious stimulus. Tissue damage and mechanical stress leads to inflammation and further to local swelling. Swelling itself is significant contributor in pain development.

Ideal pain management would attack pain development at most sites possible. The current clinical practice in the US applies a derivate of an opioid analgesic combined with acetaminophen, thereby influencing pain development at central perception by the opioid analgesic and acetaminophen and a peripheral analgesic effect of acetaminophen. The exact mechanism of the peripheral effect is not known.

This clinical practice disregards the positive effect of medications influencing the peripheral inflammatory response, namely nonsteroidal anti-inflammatory drugs (NSAIDs). NSAIDs affect pain development by blocking the synthesis of arachidonic acid metabolites, inhibiting peripheral inflammatory response and central pain perception. The major reason for not applying NSAIDs in the treatment of acute fracture pain is an experimental animal study showing decreased bone healing in relation to NSAID usage.

However, clinical data thus far is inconclusive, whether bone healing is affected in humans and whether NSAIDs should be avoided in the setting of bone fractures.

This proposed study will give an answer whether the usage of NSAIDs in acute fractures has a negative effect on bone healing.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 to < 60
* Isolated ankle fracture type SER II
* Ability to speak and understand English
* BMI< 35

Exclusion Criteria:

* ASA>3
* Previous or acute gastric bleeding
* Renal insufficiency (Creatinine: >1.27mg/dl)
* Liver insufficiency (Child-Pugh-Wert: 10-15)
* Malignant tumor
* Rheumatoid arthritis
* Heart failure (NYHA III-IV)
* High frequency absolute arrhythmia
* Patients with known psychiatric illness
* Coagulopathy
* Asthma
* Function limiting disease of the lower extremity, besides what is mentioned in the inclusion criteria
* Adults unable to consent
* Pregnant women
* Prisoners
* Workers Comp patient
* Early fracture displacement (within first 2 weeks) indicating need for surgery
* Polytrauma
* Concurrent participation in another clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
fracture healing as measured by radiographic evaluation | 12 weeks
  fracture healing at 12 weeks followup

SECONDARY OUTCOMES:
pain level improvement as measured by VAS score | 1 week, 2 weeks, 6 weeks, 9 weeks and 12 weeks
  VAS score
functional improvement as measured by AAOS score | 1 weeks, 2 weeks 6 weeks, 9 weeks and 12 weeks
  AAOS scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Steffner, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States